CLINICAL TRIAL: NCT00018122
Title: Patterns and Natural History of Insulin Secretion in Islet Cell Transplant Recipients and Controls (Project 2 of JDFI Washington University Center for Islet Transplantation, KS Polonsky, PI)
Brief Title: Patterns and Natural History of Insulin Secretion in Islet Cell Transplant Recipients and Controls
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Other Study IDs: NCRR-M01RR00036-0779
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Diabetes Mellitus
Keywords: Islet cell transplant
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This grant is to study patients that have received a kidney transplant AND an Islet Cell transplant and to discover how the transplant is functioning. We will seek to have several patients who have had a kidney transplant but do NOT have either type of diabetes. These patients will serve as the "control group" since they will also be on immunosuppressive medications but are not affected by abnormal blood sugars. This will allow investigators to develop an understanding of how these immunosuppressive medications affect glucose metabolism (blood sugar levels) and insulin utilization (how the body uses insulin).

DETAILED DESCRIPTION:
If Islet Cell transplants are to become a reasonable treatment alternative for patients with type 1 diabetes, there must be knowledge about how the islet cells function after transplant {islet cells are responsible for making the insulin the body needs in order to control blood sugar). This knowledge would allow for improvements in the islet cell transplant procedure itself, as well as possible alterations of the immunosuppressive medications (drugs that prevent rejection) that are prescribed. There are two basic kinds of diabetes, type 1 (formally known as Insulin Dependent or Juvenile diabetes) and type 2 (formally known as Adult-Onset or Non-insulin dependent) diabetes. The patients in this study will be affected by type 1 diabetes. After the transplant, it is hoped they will no longer need insulin injections. It is possible patients may need to take pioglitazone and/or metformin, however, this will be prescribed in Project 1, if needed.

The medications used for this study include: C-peptide. This is a synthetic product (not from human or animal sources) that is man-made and identical to the C-peptide made by the body. C-peptide is made at the same time as insulin, one molecule of insulin equals one molecule C-peptide. By giving C-peptide that is synthetic, researchers can measure how the C-peptide breaks down in the body, which could then be related to how insulin breaks down in the body. Somatostatin will also be used during the same test as the C-peptide. While receiving Somatostatin, the production of insulin by the patient will be stopped. This medication will only be given for 4 hours and the blood sugar will be monitored during the entire procedure. Insulin & Glucose will also be given by IV during certain tests to regulate the blood sugar. Blood sugars will be maintained within a certain level and this will be achieved through the administration of insulin and/or glucose. The patient's blood sugar will be monitored at frequent intervals throughout the various procedures.

ELIGIBILITY:
Type 1 diabetics that have received a kidney transplant as well as (under Project 1) Islet Cell Transplant. A control group of 8 kidney transplant recipients who do not have diabetes will also be sought. Age range for both groups is expected to fall in the 25-50 year/old range based upon statistical data, although those between the ages of 18 and 65 may also qualify.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States